CLINICAL TRIAL: NCT06383494
Title: GMA-Tulip, I-gel and the LMA-Supreme (LMA-S) Devices in Airway Management Under General Anesthesia, a Randomized Controlled Study (GLAM-I)
Brief Title: GMA-Tulip, I-gel and the LMA-Supreme (LMA-S) Devices in Airway Management (GLAM-I)
Acronym: GLAM-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Wang Jiangling, Principal Investigator, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-2024-356（IIT）
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia; Airway Remodeling
Keywords: Supraglottic airway device; Laryngeal inlet encapsulation; LMA-Supreme; i-gel; Fiberoptic alignment; Optimal anatomical position
MeSH Terms: conditions — Airway Remodeling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, outcome assessor and statistician were blind to the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LMA Supreme group (Active Comparator): Patient in LMA supreme group received device of LMA supreme for airway management (one of supraglottic airway device for airway management during general anesthesia)
  Interventions: Device: LMA supreme group
- I-gel group (Active Comparator): Patient in I-gel group group received device of I-gel for airway management (one of supraglottic airway device for airway management during general anesthesia)
  Interventions: Device: I-gel group
- GMA-Tulip group (Experimental): Patient in GMA-Tulip group group received device of GMA-Tulip for airway management (one of supraglottic airway device for airway management during general anesthesia)
  Interventions: Device: GMA-Tulip

INTERVENTIONS:
Device: LMA supreme group — Patient in this group received LMA supreme (one of laryngeal airway management device) for airway management during general anesthesia
  Arms: LMA Supreme group
Device: I-gel group — Patient in this group received I-gel laryngeal (one of laryngeal airway management device) for airway management during general anesthesia
  Arms: I-gel group
Device: GMA-Tulip — Patient in this group received GMA-Tulip (one of laryngeal airway management device) for airway management during general anesthesia
  Arms: GMA-Tulip group

SUMMARY:
Patients were randomly assigned to three supraglottic airway devices (SADs) groups for airway management after anesthesia induced. Fiberoptic bronchoscope (FB) guided glottic exposure grading was performed and other airway management quality was recorded.

DETAILED DESCRIPTION:
Mechanical ventilation was volume controlled and time cycled with tidal volumes (6-8 ml/kg) set to maintain peak inspiratory pressures of less than 20 cm H2O and ventilatory frequency adjusted to maintain end-tidal carbon dioxide (PETCO2) at 35-45 mmHg. Then a fiberoptic bronchoscope was passed through airway tube into the device to perform glottic exposure grading. Peak airway pressure, incidence of pharyngalgia, bleeding, hoarseness, and dysphagia were recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old;
* American Society of Anesthesiologists (ASA) I-III;
* Body mass index (BMI)<30Kg/m2;
* Scheduled for elective breast or lower abdominal surgery with an estimated duration of less than 4 hours;
* Providing written inform consent.

Exclusion Criteria:

* History of oropharyngeal surgery and anatomical abnormalities;
* Limited movement of the cervical spine;
* High risk of reflux/aspiration;
* Emergency surgery;
* Acute throat inflammation and upper respiratory infection;
* History of chronic bronchitis or asthma;
* Cognitive dysfunction and inability to communicate;
* Participating in other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Glottic exposure grading | From the insertion of supraglottic airway device to the end of surgery.
  Fiberoptic bronchoscope (FB) guided glottic exposure grading was performed.

SECONDARY OUTCOMES:
Peak inspiratory pressures | From the insertion of supraglottic airway device to 15 minutes after insertion.
  Record peak airway pressure during surgery.
Plateau inspiratory pressures | From the insertion of supraglottic airway device to 15 minutes after insertion.
  Record plateau airway pressure during surgery.
Oropharyngeal leak pressure | From the insertion of supraglottic airway device to 30 minutes after insertion
  Measure the oropharyngeal leak pressure after insertion of supraglottic airway device
Oropharyngeal leak pressure at 30 and 45 degrees of head rotation | From the insertion of supraglottic airway device to 30 minutes after insertion
  Measure the oropharyngeal leak pressure at 30 and 45 degrees of head rotation after insertion of supraglottic airway device
Ventilation quality | From the insertion of supraglottic airway device to 15 minutes after insertion
  Record the ventilation quality after the insertion of supraglottic airway device. In specific, The Ventilation Quality Score consists of three components: presence of normal CO₂ waveform, bilateral symmetrical chest rise, and absence of air leak at 20 mmHg airway pressure. Total scores range 0-3, with 0 indicating poor ventilation quality and 3 representing optimal ventilation.
Abnormally ventilation events during surgery | From the insertion of supraglottic airway device to the end of surgery
  Record the abnormally ventilation events (air leakage, abnormal carbon dioxide wave, higher airway pressure, hypoxemia, supraglottic airway device adjustment, change into intubation) during surgery
Side effects at the end of surgery | From the insertion of supraglottic airway device to the patient's transfer to the ward. An average of 3 hours.
  Record side effects (blooding on the supraglottic airway device, pharyngalgia, hoarseness) at the end of surgery.
Side effects and adverse events 24 hours after surgery | Postoperative day 1.
  Record side effects (pharyngalgia, hoarseness, cough when drinking), and adverse events (pneumonia, hypoxemia) 24 hours after surgery.
Nasogastric tube insertion success rate | From the initial insertion to the successful placement of nasogastric tube. An average of 20 minutes.
  Record the nasogastric tube insertion success rate
Nasogastric tube insertion attempts | From the initial supraglottic airway device insertion to the successful placement of nasogastric tube. An average of 20 minutes.
  Record the number of attempts for nasogastric tube insertion
Nasogastric tube insertion time | From the initial supraglottic airway device insertion to the successful placement of nasogastric tube. An average of 20 minutes.
  Record the duration (seconds from insertion initiation to successful placement) of nasogastric tube insertion
Nasogastric tube insertion difficulty | From the initial supraglottic airway device insertion to the successful placement of nasogastric tube. An average of 20 minutes.
  Record the insertion difficulty (1-3 scale; 1=easy, 3=difficult) of nasogastric tube placement
Reflux or aspiration risk | From the insertion of s SAD to the end of surgery. An average of 3 hours.
  Record gas/fluid volume during the surgery
Supraglottic airway device insertion duration | From the mouth open to the device seated upon encountering resistance, averaging approximately 10 seconds.
  Record the insertion duration (seconds from insertion initiation to successful placement) of SADs
Supraglottic airway device insertion difficult | From the mouth open to the device seated upon encountering resistance, averaging approximately 10 seconds.
  Record the insertion difficulty (1-3 scale; 1=easy, 3=difficult) of SADs
Supraglottic airway device insertion times | From the mouth open to the device seated upon encountering resistance or able to ventilation after device's adjustment/reinsertion, averaging approximately 10 seconds.
  Record the number of SAD insertion attempts.

CONTACTS AND LOCATIONS:
Overall Officials: Jiangling Wang, Ph. D, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China